CLINICAL TRIAL: NCT01547130
Title: A Single Blind, Parallel Group, Randomized Controlled Trial Comparing Solution PEG Based Colon Preparation (HalfLytely) Versus Bolus Luke Warm Saline (Shudh) and Yoga Exercise for Large Bowel Cleansing Prior to Colonoscopy
Brief Title: Yoga and Bolus Lukewarm Saline as Rapid Colonoscopy Preparation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arya, Vijaypal, M.D., P.C. (Individual)
Responsible Party: Principal Investigator, Vijaypal Arya MD, FACP, FACG, AGAF., Associate Director, Endoscopy, Arya, Vijaypal, M.D., P.C.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WHMC-2008-35
Record Dates: First submitted 2012-02-26; First posted 2012-03-07 (Estimated); Results first posted 2015-03-04 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-02

CONDITIONS: Colonic Neoplasms
Keywords: Colonoscopy; Yoga; Complementary and alternative medicine; Bowel cleansing; Large bowel preparation; Cancer screening; Colorectal cancer
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BLS and Yoga exercise (Active Comparator): Patients will take a bolus intake of 8 oz. (240mL) to 16 oz. (480mL) of lukewarm saline water and perform yoga poses.
  Interventions: Drug: Normal (0.9%) saline
- PEG (HalfLytely) (Active Comparator): Patients followed the preparation method according to the manufacturer's standard instructions.
  Interventions: Drug: HalfLytely

INTERVENTIONS:
Drug: Normal (0.9%) saline — A total of 2L solution at lukewarm temperature (37.2-38.8 degrees Centigrade)consumed as bolus intake (8-16 oz in one to two minutes) alternating with yoga exercises.
  Arms: BLS and Yoga exercise
Drug: HalfLytely — A total of 2L solution prepared as per manufacturers instructions and sipped until bowel movements are clear.
  Arms: PEG (HalfLytely)

SUMMARY:
A quality colonoscopy examination remains as the gold standard for colorectal cancer screening, but effective large bowel cleansing prior to colonoscopy is still not achieved in all cases that undergo the procedure. Currently, the most widely used cleansing methods employ balanced electrolyte-polyethylene glycol (PEG) solutions. However, a very large volume of PEG solution is required for it to be effective, and many patients refuse to drink a sufficient amount due to non-palatability. In this study, the investigators compare a novel colon preparation method--bolus lukewarm saline with yoga exercise--with a PEG based solution (HalfLytely) for large bowel cleansing.

DETAILED DESCRIPTION:
Effective large bowel cleansing prior to colonoscopy is still not achieved in all cases that undergo the procedure. The use of balanced electrolyte-polyethylene glycol (PEG) solution have improved the cleansing results and shortened the time needed for preparing the bowel. The problem with using PEG solution alone is the relatively large volume of the solution that the patients need to drink. The recommendation is to drink the solution until diarrhea fluid is clear and often 4 L or more is needed. Many patients refuse to drink the sufficient volume needed to get a clean colon due to non-palatability. Good results of bowel cleansing have also been reported with sodium phosphate solution or tablets.

The fluid volume needed to drink along with sodium phosphate is generally no problem but this regimen causes electrolyte disturbances and renal insufficiency that usually are subclinical and of no significance. Several combinations of PEG solution and laxatives have been tested before. Low-volume PEG plus Bisacodyl preparation was better tolerated but it was not as effective as standard large-volume PEG and associated with abdominal cramping.

PEG solution 2L and Bisacodyl is used for large bowel cleansing in many centers in the United States and is the standard regimen used in our colonoscopy unit. In this study the investigators compare this standard regimen taken day before colonoscopy with Bolus lukewarm saline solution taken orally with yoga exercise on the day of colonoscopy.

The result of large bowel cleansing is evaluated during the colonoscopy according to a validated scoring method. Time to the first bowel movement and total preparation time are compared. Solution palatability, patient acceptability, abdominal symptoms, discomfort and subjective grading of how hard/easy it was to complete the cleansing program are evaluated with questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled to undergo elective complete colonoscopy as an outpatient.
* Aged 18 or older.
* The patient gives written informed consent and can understand the information given.
* The patient can participate in the study only once.

Exclusion Criteria:

* Sodium chloride sensitivity.
* Limitation to exercise.
* Earlier resection of the large bowel or rectum.
* Known active colitis.
* Ileus or gastrointestinal obstruction.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2008-05; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vijaypal Arya, MD, Principal Investigator — Wyckoff Heights Medical Center
Locations (1):
- Vikalp Inc., Middle Village, New York, United States

REFERENCES:
- [Derived] Arya V, Gupta KA, Valluri A, Arya SV, Lesser ML. Rapid colonoscopy preparation using bolus lukewarm saline combined with sequential posture changes: a randomized controlled trial. Dig Dis Sci. 2013 Aug;58(8):2156-66. doi: 10.1007/s10620-013-2598-9. Epub 2013 Mar 2. PMID 23456498

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, single-center, single-blinded (to the endoscopists) and active-control study. Patients undergoing elective colonoscopy between May 2008 and December 2010 were recruited. Location: Medical Clinic.
Pre-assignment Details: No events were recorded. None of the enrolled participants were excluded from the trial before assignment to groups. However, 14 no show ups for procedure were identified.
Groups:
- Shudh Colon Cleanse (SCC) Group: Patients will take a bolus intake of 8 oz. (240mL) to 16 oz. (480mL) of lukewarm saline water and perform yoga poses.
- HalfLytely Colon Prep (HCP): Patients followed the preparation method according to the manufacturer's standard instructions.
Period: Overall Study
Arm/Group | Shudh Colon Cleanse (SCC) Group | HalfLytely Colon Prep (HCP)
Started | 74 | 73
Completed | 65 | 68
Not Completed | 9 | 5
Not completed — Lost to Follow-up | 9 | 5

BASELINE CHARACTERISTICS:
Groups:
- HalfLytely Colon Prep (HCP) Group: Patients followed the preparation method according to the manufacturer's standard instructions.
- Total: Total of all reporting groups
Arm/Group | Shudh Colon Cleanse (SCC) Group | HalfLytely Colon Prep (HCP) Group | Total
Number analyzed (Participants) | 74 | 73 | 147
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 72 | 73 | 145
  >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (10.5) | 44.8 (10) | 44.2 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 43 | 91
  Male | 26 | 30 | 56
Region of Enrollment [Number; unit: participants]
  United States | 74 | 73 | 147

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Large Bowel Cleansing as Assessed by the Physician Performing the Colonoscopy
Description: The primary endpoint was the "success" rate of the preparations. Preparation efficacy was evaluated by a single, blinded endoscopist (V.A.), who performed all of the colonoscopies. The evaluation involved the rating of six anatomical segments of the colon (rectum, sigmoid, descending colon, transverse colon, ascending colon and cecum) on the 5 point Arya Bowel Prep Scale (ABPS). Aggregating the segmental scores resulted in overall scores. Grade A was defined as a total overall score of 19-24, grade B as a score of 13-18, grade C as a score of 7-12, and grade D as a score of 0-6. Grade A or B preparation was considered "successes", while grade C or D was considered "failures." To assess the reliability of ABPS, we trained 4 gastroenterologists and 3 fellows.
Time Frame: Within 48 hours of bowel preparation
Population: The non-inferiority margin was set at -15%. This means the intervention will be considered non-inferior if the difference in success rates is less than 15%. The study was designed to have 90% power to establish non-inferiority when the two treatment groups are equivalent using a one-tailed test at the 5% significance level.
Measure: Mean (Standard Deviation); unit: Score
Groups:
- Shudh Colon Cleanse (SCC) Group: Yoga contained a 32-oz plastic pitcher and 9-gm salt sachets (Iodine-free table salt - USP grade sodium chloride) for preparation of 0.9% saline (1 sachet in 32-oz lukewarm water (37.2-38.8 degrees Centigrade or 99-102 degrees Fahrenheit)), an instructional leaflet, and a DVD providing instructions of the bowel preparation process. Patients were instructed to fill the pitcher with 16-oz of hot water and 16-oz of room temperature water to reach the lukewarm temperature. Patients could add a twist of lemon if the solution was unpalatable to them.
- HalfLytely Colon Prep (HCP) Group: Patients in the HCP group followed the preparation method according to the manufacturer's standard instructions. Patients were instructed to stay on clear liquids the entire day before the colonoscopy. Two tablets of bisacodyl delayed-release tablets with water were taken at around 1:00 pm. Patients were instructed to start drinking the solution after a bowel movement or around 7 pm if no bowel activity occurred. They were instructed to sip all of the solution at a rate of 8 oz. every 10 minutes.
Arm/Group | Shudh Colon Cleanse (SCC) Group | HalfLytely Colon Prep (HCP) Group
Number analyzed (Participants) | 65 | 68
Score | 18.69 (5.34) | 20.1 (3.51)

2. Secondary Outcome: Palatability of Bowel Prep
Description: Patients completed a symptom questionnaire where they rated solution palatability of their assigned prep on a 1-5 Likert scale. A rating of more than 3 was considered as "Palatable".
Time Frame: Upto 24 weeks
Population: All subjects enrolled and completed the bowel preparation. .
Measure: Number; unit: participants
Groups:
- Shudh Colon Cleanse (SCC) Group: Solution palatability of SCC by subjects based on 1-5 scale (1-not palatable and 5-Palatable). A questionnaire was used to collect the data.
- HalfLytely Colon Prep (HCP) Group: Solution palatability of HCP by subjects based on 1-5 scale (1-not palatable and 5-Palatable). A questionnaire was used to collect the data.
Arm/Group | Shudh Colon Cleanse (SCC) Group | HalfLytely Colon Prep (HCP) Group
Number analyzed (Participants) | 65 | 68
participants | 48 | 38

3. Secondary Outcome: Subjective Grading by Patients on Willingness to Repeat the Large Bowel Preparation.
Description: Subjects rated the SCC as "Willingness to repeat the same prep in future"
Time Frame: Upto 24 weeks
Population: Patients completed a questionnaire where they rated willingness to repeat the preps on a 1-5 Likert scale.
Measure: Number; unit: participants
Groups:
- Shudh Colon Cleanse (SCC) Group: Subjects rated the SCC as palatable
- HalfLytely Colon Prep (HCP) Group: Subjects rated the HCP as palatable
Arm/Group | Shudh Colon Cleanse (SCC) Group | HalfLytely Colon Prep (HCP) Group
Number analyzed (Participants) | 65 | 68
participants | 44 | 40

4. Secondary Outcome: Patient-reported Adverse Events.
Description: Patients from both groups reported adverse events in a symptom questionnaire.
Time Frame: Upto 24 weeks
Population: Patients from both groups reported adverse events in a symptom questionnaire.
Measure: Number; unit: participants
Groups:
- Shudh Colon Cleanse (SCC) Group: Patients take a bolus intake of 8 oz. (240mL) to 16 oz. (480mL) of lukewarm saline water and perform yoga poses. Adverse events were recorded on questionnaire.
- HalfLytely Colon Prep (HCP) Group: Patients followed the preparation method according to the manufacturer's standard instructions. Subjects recorded adverse events.
Arm/Group | Shudh Colon Cleanse (SCC) Group | HalfLytely Colon Prep (HCP) Group
Number analyzed (Participants) | 65 | 68
participants | 32 | 46

5. Secondary Outcome: Total Preparation Time
Description: Patients in both groups were provided with a questionnaire to record the total time required from start of assigned prep to completion of the prep.
Time Frame: Upto 24 weeks
Population: Patients in both groups were provided with a questionnaire to record the total time required from start of assigned prep to completion of the prep.
Measure: Mean (Full Range); unit: hours
Arm/Group | Shudh Colon Cleanse (SCC) Group | HalfLytely Colon Prep (HCP) Group
Number analyzed (Participants) | 65 | 68
hours | 1.9 [1.25 to 4] | 10.9 [4 to 18]

ADVERSE EVENTS:
Time Frame: Same day
Arm/Group | Shudh Colon Cleanse (SCC) Group | HalfLytely Colon Prep (HCP) Group
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/68
Other Adverse Events (participants affected / at risk) | 25/65 | 28/68
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Shudh Colon Cleanse (SCC) Group (N=65) | HalfLytely Colon Prep (HCP) Group (N=68)
Nausea (Gastrointestinal disorders) | 25 | 28
Vomiting (Gastrointestinal disorders) | 3 | 12

LIMITATIONS AND CAVEATS:
Shudh Colon Cleanse (SCC) is suitable to only 30% of patients who are undergoing colonoscopy. A multi-center study is warranted to confirm these results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No